CLINICAL TRIAL: NCT02415530
Title: Early Family-Based Intervention for Developmental Enforcement of Premature Infants
Brief Title: Early Family Based Intervention in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul St. Mary's Hospital (Other); CHA University (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1501097642
Record Dates: First submitted 2015-04-05; First posted 2015-04-14 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Very Low Birth Weight Infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Term infant control (Placebo Comparator): term infant without intervention
  Interventions: Other: No intervention
- VLBW infant control (Placebo Comparator): very low birth weight infant without intervention
  Interventions: Other: No intervention
- VLBW infant intervention (Experimental): Combined home visiting and group intervention for very low birth weight infant
  Interventions: Behavioral: Combined home visiting and group intervention

INTERVENTIONS:
Behavioral: Combined home visiting and group intervention — home visit includes pre-discharge meeting with parents; education of appropriate feeding, breastfeeding, sleeping, position of baby, defecation, environment for baby care and resuscitation on emergency situation first visit (5 days after discharge); understanding baby's sign check feeding, sleeping, sanitation, defecation, environment second visit (14 days after discharge); understanding baby's sign and baby's development support parents check feeding, sleeping, sanitation, defecation, environment special situation third visit (4 weeks after discharge) understanding baby's sign and baby's development support parents special situation fourth visit (8 weeks after discharge) same as third visit Group intervention for parental support with baby 12 times during corrected age 3~6 months
  Arms: VLBW infant intervention
Other: No intervention — No intervention
  Arms: Term infant control; VLBW infant control

SUMMARY:
This is randomized controlled trial investigating the effect of early intervention in very low birth weight infants after discharge from NICU on neurodevelopmental outcome. Other than control group of VLBW infants, study population includes term infants to compare neurodevelopmental outcome.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants < 32 weeks of gestation or 1,500 gm of birth weight
* normal term infants

Exclusion Criteria:

* major congenital anomaly
* neuromuscular disease
* chromosomal anomaly
* triplets or more multiplets

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development III, mental developmental index | Corrected age 10 months

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development III, psychomotor developmental index | Corrected age 10 month
CES-D-depression screening tool | Corrected age 2 month & 6 month
Maternal attachment | Corrected age 2 month & 6 month
Temperament scale | Corrected age 8 month
Wechsler Intelligence Scale | 8 years of age
Conners ADHD/DSM-IV Scales | 8 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Ee-kyung Kim, Principal Investigator — Seoun National University Hospital
Locations (3):
- South Korea (3):
  - CHA Gangnam Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul